CLINICAL TRIAL: NCT03431090
Title: HAPLEUK17, Haploidentical Hematopoietic Cell Transplantation for Children With Hematologic Malignancies and Myelodysplasia
Brief Title: Haploidentical Hematopoietic Cell Transplantation for Children With Hematologic Malignancies and Myelodysplasia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-00516
Record Dates: First submitted 2017-12-27; First posted 2018-02-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Myelodysplasia; Hematologic Malignancy
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: The mobilized peripheral blood cell collection (apheresis product) will be processed using a Miltenyi CliniMACS device according to the manufacturing instructions. The processing will deplete the αβTCR+ cells and CD19+ cells from the apheresis product to formulate the graft.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CliniMACS Isolation (Experimental): The mobilized peripheral blood cell collection (apheresis product) will be processed using a Miltenyi CliniMACS device according to the manufacturing instructions. The processing will deplete the αβTCR+ cells and CD19+ cells from the apheresis product to formulate the graft.
  Interventions: Device: CliniMACS® TCRαβ/CD19 Combined Depletion System

INTERVENTIONS:
Device: CliniMACS® TCRαβ/CD19 Combined Depletion System — The mobilized peripheral blood cell collection (apheresis product) will be processed using a Miltenyi CliniMACS device according to the manufacturing instructions. The processing will deplete the αβTCR+ cells and CD19+ cells from the apheresis product to formulate the graft.

SUMMARY:
This is a Phase I/II study designed to evaluate the kinetics of hematopoietic reconstitution and the incidence of acute chronic GVHD after partially matched related donor hematopoietic cell transplantation using an αβTCR/CD19+ cell depleted graft.

DETAILED DESCRIPTION:
Less than 30% of patients undergoing hematopoietic cell transplantation (HCT) will have an HLA-matched sibling donor. There is a high likelihood of being unable to identify a perfect HLA matched unrelated donor, and the time to procure the marrow if such a donor is available is generally >3 months. An emerging body of literature suggests that related haploidentical HCT with innovative graft engineering may provide equal, or possibly superior, outcomes to conventional unrelated donors. This protocol is designed to test the hypothesis that HCT using an αβT cell / CD19+ B cell depleted graft from partially matched related donors will result in rapid, durable hematopoietic engraftment and rapid immune reconstitution with an acceptably low risk of severe acute and chronic GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Patient lacks an HLA matched sibling donor.
* Meets criteria nonhematopoietic organ function according to NCH BMT SOP09.
* If subjects have received a first HCT, they must be eligible for a second HCT if their disease has recurred.
* High resolution HLA and KIR typing
* The subject cannot have an active untreated infection. Viremia by PCR analysis is not considered an active infection but may require immediate viral prophylaxis. Patients with possible fungal infections must have had at least 2 weeks of appropriate anti- fungal therapy and be asymptomatic.
* Negative pregnancy test for females ≥11 years of age or post- menarche.
* Sexually active males and females of childbearing potential must agree to use a form of contraception considered effective and medically acceptable by the Investigator. (Non-childbearing potential defined as pre-menarche, greater than one year post-menopausal or surgically sterilized).
* Subjects must be ≤30 years at the time of consent.
* Signed consent by parent/guardian and assent if appropriate for subjects < 18 years of age. Signed consent by patient/subject if ≥18 years of age.

Exclusion Criteria:

* Patient does not have a suitable donor who is willing and able (meets donor criteria).
* Patient has donor-specific anti-HLA antibodies at the time of enrollment
* Patient reports a history of allergic reactions to murine protein

Donor Eligibility:

* The donor must be ≥18 years of age at the time of the informed consent conference.
* The donor must be a related donor
* The donor will be evaluated according to the current NCH BMT SOP 04 and must meet all criteria.
* The donor must be able and willing to undergo G-CSF mobilization and stem cell apheresis.
* The patient does not have donor specific anti-HLA antibodies

Max Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Measure rates of neutrophil and platelet engraftment | 4 years
  Patients undergoing partially matched related donor hematopoietic cell transplantation with an αβT cell / CD19+ B cell depleted graft should have an improved rate of engraftment.
Measure incidence of acute GVHD | 4 years
  Patients undergoing partially matched related donor hematopoietic cell transplantation with an αβT cell / CD19+ B cell depleted graft should have a lower incidence of acute and chronic GVHD.
Measure rates of immune reconstitution | 4 years
  Patients undergoing partially matched related donor hematopoietic cell transplantation with an αβT cell / CD19+ B cell depleted graft should have a improved rate of immune reconstitution.
Measure rates of platelet engraftment | 4 years
  Patients undergoing partially matched related donor hematopoietic cell transplantation with an αβT cell / CD19+ B cell depleted graft should have an improved rate of engraftment.
Measure incidence of chronic GVHD | 4 years
  Patients undergoing partially matched related donor hematopoietic cell transplantation with an αβT cell / CD19+ B cell depleted graft should have a lower incidence of acute GVHD.

SECONDARY OUTCOMES:
Measure overall survival | 4 years
  Patients undergoing partially matched related donor hematopoietic cell transplantation with an αβT cell / CD19+ B cell depleted graft overall survival and relapse rate/disease free survival rates will be evaluated as compared to other treatment methodologies.
Define nonhematopoietic regimen related toxicities | 4 years
  Patients undergoing partially matched related donor hematopoietic cell transplantation with an αβT cell / CD19+ B cell depleted graft will be evaluated for nonhematopoietic regimen related toxicities.
Measure relapse rate | 4 years
  Patients undergoing partially matched related donor hematopoietic cell transplantation with an αβT cell / CD19+ B cell depleted graft overall survival
Measure disease free survival | 4 years
  Patients undergoing partially matched related donor hematopoietic cell transplantation with an αβT cell / CD19+ B cell depleted graft overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No